CLINICAL TRIAL: NCT03373006
Title: A Phase II Study to Evaluate Axumin PET/CT for Risk Stratification for Laser Focal Therapy of Intermediate Risk Localized Prostate Cancer
Brief Title: A Phase II Study to Evaluate Axumin PET/CT for Risk Stratification for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HALO Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DMI Axumin-001; Protocol. No: 20171334 (Other: Western IRB (WIRB)); Study No: 1176339 (Other: Western IRB (WIRB))
Record Dates: First submitted 2017-12-08; First posted 2017-12-14 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Cohort
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Men with Gleason Score 7 prostate cancer (Experimental): Men seeking focal therapy for Gleason Score 7 prostate cancer will receive Axumin PET/CT imaging to detect metastasis which will result in exclusion from laser focal therapy.
  Interventions: Drug: Axumin PET/CT

INTERVENTIONS:
Drug: Axumin PET/CT — Synthetic amino acid uptake agent injection followed by imaging
  Other Names: PET/CT scan

SUMMARY:
To investigate the utility of fluciclovine F 18 for evaluation for metastatic disease in men undergoing laser focal therapy of prostate cancer and the impact on inclusion for a focal therapy cohort.

DETAILED DESCRIPTION:
DESCRIPTION OF DRUG

Mechanism of action:

Fluciclovine F 18 is a synthetic amino acid transported across mammalian cell membranes by amino acid transporters, such as LAT-1 and ASCT2, which are upregulated in prostate cancer cells. Fluciclovine F 18 is taken up to a greater extent in prostate cancer cells compared with surrounding normal tissues.

Pharmacodynamics:

Following intravenous administration, the tumor-to-normal tissue contrast is highest between 4 and 10 minutes after injection, with a 61% reduction in mean tumor uptake at 90 minutes after injection.

Pharmacokinetics:

Distribution: Following intravenous administration, fluciclovine F 18 distributes to the liver (14% of administered activity), pancreas (3%), lung (7%), red bone marrow (12%) and myocardium (4%). With increasing time, fluciclovine F 18 distributes to skeletal muscle.

Excretion: Across the first four hours post-injection, 3% of administered radioactivity was excreted in the urine. Across the first 24 hours post-injection, 5% of administered radioactivity was excreted in the urine.

TEST PRODUCT, DOSE, AND ROUTE OF ADMINISTRATION All subjects will receive a single IV dose of 10mCi (370MBq) +20%18F-fluciclovine immediately prior to PET scan.

Administration: Prior to PET/CT, 10mCi ±20% of 18F-fluciclovine will be administered as an IV bolus injection followed by a 10 mL saline flush, with the subject lying in a supine position. The dose will be injected into an antecubital vein or another vein that will provide access. The administration site will be evaluated pre- and post- administration for any reaction (e.g. bleeding, hematoma, redness, or infection). Documentation of administration to a subject will be recorded according to standard of care, including start of administration, injection site, date, prescription number, total volume and total radioactivity.

Packaging, Labeling and ordering: Fluciclovine F 18 is supplied as a unit dose for injection in a syringe with a radioactive concentration at a reference date and time that is stated on the container label. Each syringe is supplied in a container providing appropriate radiation shielding. Information will be provided with the shipment giving the confirmation number, radioactive concentration of injection (mCi/mL) at a stated time and date, shelf life information, protocol number and a unique prescription number. The radiochemical purity of 18F-fluciclovine injection is not less than 95% during the shelf life of the product. The order for a specific patient at a specific date and time must be made to PETNET Solutions Centralized Scheduling Team (Tel: 1 877 473 8638) and will be delivered from the radiopharmacy to the imaging site by courier. Indian Wells PET/CT Center will keep records of all shipments of fluciclovine F 18 received, dispensing and disposal/destruction performed on site in accordance with ACR and NCRP guidelines.

Imaging protocol.

1. The recommended dose is 370 MBq (10 mCi) administered as an intravenous bolus injection.
2. Begin PET scanning 3 to 5 minutes after completion of the Axumin injection
3. Proximal thigh to skull base x 5min/bed position caudocranial direction
4. Recon: Iterative
5. Iterations - 2, Subsets - 8
6. Filter Gaussian

Image interpretation: Image interpretation will be based on guidelines outlined in and derived from an international 18F-fluciclovine Reader Consensus Meeting held in June 2014 (see References) and will follow processes similar to those outlined on the on-line Axumin™ (fluciclovine F 18) Image Interpretation Training (http://jnm.snmjournals.org/content/58/10/1596.long) . Reader has undergone training in interpretation of 18F- fluciclovine PET/CT scans, and has a training set available for reference.

1. Non-Significant Risk Study Desert Positron Imaging has identified this investigation as a Non-Significant Risk (NSR) study.

PRELIMINARY WORK

1. CLINICAL STUDIES: The safety and efficacy of Axumin were evaluated in two studies (Study 1 and Study 2) in men with suspected recurrence of prostate cancer based on rising PSA levels following radical prostatectomy and/or radiotherapy.

Study 1 evaluated 105 Axumin scans in comparison to histopathology obtained by biopsy of the prostate bed and biopsies of lesions suspicious by imaging. PET/CT imaging generally included the abdomen and pelvic regions. The Axumin images were originally read by on-site readers. The images were subsequently read by three blinded independent readers. Table 4 of the package insert for Axumin shows the performance of Axumin in the detection of recurrence in each patient scan and, specifically, within the prostate bed and extra-prostatic regions, respectively. The results of the independent read were generally consistent with one another and confirmed the results of the on-site reads.

In general, patients with negative scans had lower PSA values than those with positive scans. The detection rate (number with positive scans/total scanned) for patients with a PSA value of less than or equal to 1.78 ng/mL (1st PSA quartile) was 15/25, of which 11 were histologically confirmed as positive. In the remaining three PSA quartiles, the detection rate was 71/74, of which 58 were histologically confirmed. Among the 25 patients in the first PSA quartile, there were 4 false positive scans and 1 false negative scan. For the 74 patients with PSA levels greater than 1.78 ng/mL, there were 13 false positive scans and no false negative scans. Study 2 evaluated the concordance between 96 Axumin and C11 choline scans in patients with median PSA value of 1.44 ng/mL (interquartile range = 0.78 to 2.8 ng/mL). The C11 choline scans were read by on-site readers. The Axumin scans were read by the same three blinded independent readers used for Study 1. The agreement values between the Axumin and C11 choline reads were 61%, 67% and 77%, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 45 years of age or older.
2. Diagnosis of prostate adenocarcinoma.
3. Clinical stage T1a, T1b, T1c, T2a, T2b orT2c.
4. Gleason score of 7 (3+4 or 4+3).
5. PSA density less than 0.375.
6. One, two, or three tumor suspicious regions identified on multiparametric MRI.
7. Negative radiographic indication of extra-capsular extent.
8. Karnofsky performance status of at least 70.
9. Estimated survival of 5 years or greater, as determined by treating physician.
10. Tolerance for anesthesia/sedation.
11. Ability to give informed consent.

Exclusion Criteria:

1. Presence of any condition (e.g., metal implant, shrapnel) not compatible with MRI.
2. Severe lower urinary tract symptoms as measured by an International Prostate Symptom Score (IPSS) of 20 or greater. ( (http://www.urospec.com/uro/Forms/ipss.pdf)
3. History of other Primary non-skin malignancy within previous three years.
4. Diabetes.
5. Smoker.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with Gleason 7 prostate cancer (3+4 or 4+3)
Enrollment: 20 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Feller, MD, Principal Investigator — Medical Director, Radiation Safety Officer; Bernadette M Greenwood, MSc., Study Director — Chief Research Officer
Locations (1):
- Desert Medical Imaging, Indian Wells, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Present at scientific meetings as anonymized data, anonymize reports for case studies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within one year of completing of patient #20.
Access Criteria: Attendees at CME courses and researchers visiting Desert Medical Imaging may view data from our spreasdsheets and PACS. Case reports and anonymized data will be shared at scientific meetings.

REFERENCES:
- [Background] Nanni C, Schiavina R, Brunocilla E, Boschi S, Borghesi M, Zanoni L, Pettinato C, Martorana G, Fanti S. 18F-Fluciclovine PET/CT for the Detection of Prostate Cancer Relapse: A Comparison to 11C-Choline PET/CT. Clin Nucl Med. 2015 Aug;40(8):e386-91. doi: 10.1097/RLU.0000000000000849. PMID 26053708
- [Background] Schreibmann E, Schuster DM, Rossi PJ, Shelton J, Cooper S, Jani AB. Image Guided Planning for Prostate Carcinomas With Incorporation of Anti-3-[18F]FACBC (Fluciclovine) Positron Emission Tomography: Workflow and Initial Findings From a Randomized Trial. Int J Radiat Oncol Biol Phys. 2016 Sep 1;96(1):206-13. doi: 10.1016/j.ijrobp.2016.04.023. Epub 2016 Apr 30. PMID 27511856
- [Background] Jambor I, Kuisma A, Kahkonen E, Kemppainen J, Merisaari H, Eskola O, Teuho J, Perez IM, Pesola M, Aronen HJ, Bostrom PJ, Taimen P, Minn H. Prospective evaluation of 18F-FACBC PET/CT and PET/MRI versus multiparametric MRI in intermediate- to high-risk prostate cancer patients (FLUCIPRO trial). Eur J Nucl Med Mol Imaging. 2018 Mar;45(3):355-364. doi: 10.1007/s00259-017-3875-1. Epub 2017 Nov 16. PMID 29147764
- [Background] Zarzour JG, Galgano S, McConathy J, Thomas JV, Rais-Bahrami S. Lymph node imaging in initial staging of prostate cancer: An overview and update. World J Radiol. 2017 Oct 28;9(10):389-399. doi: 10.4329/wjr.v9.i10.389. PMID 29104741
- [Background] Miller MP, Kostakoglu L, Pryma D, Yu JQ, Chau A, Perlman E, Clarke B, Rosen D, Ward P. Reader Training for the Restaging of Biochemically Recurrent Prostate Cancer Using 18F-Fluciclovine PET/CT. J Nucl Med. 2017 Oct;58(10):1596-1602. doi: 10.2967/jnumed.116.188375. Epub 2017 Apr 6. PMID 28385791

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Men With Gleason Score 7 Prostate Cancer
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Men with intermediate risk prostate cancer considering laser focal therapy
Arm/Group | Men With Gleason Score 7 Prostate Cancer
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Only males. Prostate Cancer study.
  Participants
    Female | 0
    Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20
Males over 45 with GS 3+4 or 4+3 prostate cancer [Count of Participants; unit: Participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Detection of Metastases
Description: Number of patients with detection of metastasis
  Secondary Outcome Measure Description: Number of patients with local uptake of Axumin
Time Frame: One day
Population: Patients with intermediate risk prostate cancer
Measure: Count of Participants; unit: Participants
Groups:
- Axumin Arm: Men over 45 years of age with Gleason 3+4 or 4+3 prostate cancer
Arm/Group | Axumin Arm
Number analyzed (Participants) | 20
Participants
  Participants with no detection of metastasis or local uptake | 7
  Participants with local uptake only | 8
  Participants with detection of metastasis and local uptake (1 mediastinal node and 1 osseous) | 2
  Participants with detection elsewhere and local uptake | 0
  Participants with uptake elsewhere only (thyroid) | 1
  Participants with metastasis only | 1
  Participants with uptake elsewhere only | 1
  Participants with uptake detected elsewhere and metastasis | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Patients were instructed to contact our physicians if they experienced any unexpected symptoms after their examination.
Groups:
- Men With Gleason Score 7 Prostate Cancer: Men seeking focal therapy for Gleason Score 7 prostate cancer will receive Axumin PET/CT imaging to detect metastasis which will result in exclusion from laser focal therapy.
  Axumin PET/CT: Synthetic amino acid uptake agent injection followed by imaging
  No adverse events were observed.
Arm/Group | Men With Gleason Score 7 Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
One limitation of this study was the mall sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT03373006/Prot_002.pdf
  • Informed Consent Form (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT03373006/ICF_001.pdf